CLINICAL TRIAL: NCT00558506
Title: Pilot Open Label Clinical Trial With Abatacept in Ankylosing Spondylitis
Acronym: Aba-AS-01
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABATACEPT-AS-01
Record Dates: First submitted 2007-11-14; First posted 2007-11-15 (Estimated); Last update posted 2008-02-26 (Estimated); Status verified 2007-09

CONDITIONS: Ankylosing Spondylitis
Keywords: Ankylosing spondylitis; activity; treatment; clinical trial
MeSH Terms: conditions — Spondylitis, Ankylosing; Motor Activity | interventions — Abatacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Abatacept
  Interventions: Drug: abatacept

INTERVENTIONS:
Drug: abatacept — intravenously 750mg (in patients with weight of 60- 100kg)

SUMMARY:
This is an open-label trial investigating the efficacy and safety of abatacept in ankylosing spondylitis. It is planned to treat 30 patients with ankylosing spondylitis from baseline up to week 30. Abatacept will be administered intravenously according to the prescription used in rheumatoid arthritis.

DETAILED DESCRIPTION:
Clinical manifestations and prevalence of ankylosing spondylitisAnkylosing spondylitis (AS) is a chronic inflammatory disease which affects primarily the spine and the sacroiliac joints, but extraspinal structures such as peripheral joints, the enthesis (insertion of tendons/ligaments at bone), the eye (uveitis) and the aorta can also be involved. There is a strong association between AS and the MHC class I antigen HLA-B27 which is positive in 90-95% of patients. About 5% of HLA-B27-positve individuals do develop ankylosing spondylitis during lifetime, starting in more than 95% at an age younger than 45 years. The overall prevalence of AS has been estimated to be between 0.2 and 1.2%. These differences can mainly be explained by differences in the HLA-B27 prevalence in different populations. Current treatment of ankylosing spondylitisRecent ASAS/EULAR recommendations for the treatment of AS state that for the predominant axial manifestations there are only two groups of effective drugs: the NSAIDs and, more recently, the TNF-blockers 1. Thus, in contrast to rheumatoid arthritis and other inflammatory rheumatic diseases such as SLE treatment with DMARDs does not play a role in the mangement of AS. Most recently, we could show in three open label studies that drugs such as leflunomide2, the IL-RA anakinra3 and methotrexate 4 are not effective in AS. Sulfasalazine, the DMARD most often used for the treatment of AS, has, if at all, also only a very limited efficacy. About 20-30% of AS patients have been estimated to be potential candidates for treatment with TNF-blockers because their disease is still active despite an adequate therapy with NSAIDs. From the AS patients treated with TNF-blockers, about 50% show a 50% improvement in their disease acitivity (BASDAI), but 50% do not. Especially for the latter patients with no or only a suboptimal response to anti-TNF agents alternative treatment options are urgently needed. Evidence for ankylosing spondylitis as an autoimmune disease and thepotential role of T cells in the pathogenesisWe have argued already 10 years ago that autoimmunity plays an important role in the pathogenesis of ankylosing spondylitis (AS). Although there is no direct evidence, as in nearly all 'suspected' autoimmune diseases, of an autoimmune response in AS it has been proposed repeatedly over the last years that the cartilage is the most likely target of an autoimmune response in AS. Histological studies and magnet resonance imaging investigations suggest that the primary site of inflammation is the cartilage/bone interphase. Mononuclear cell infiltrates are mainly found in cartilage and the subchondral bone. In early and active sacroiliitis, T cells and macrophages are dominant in these infiltrates underlining the relevance of a specific cellular immune response . This was further backed by recent studies from our group demonstrating mononuclear infiltrates (including both CD4+ and CD8+ T cells) of cartilage by investigating femoral heads and facette joints (small joints of the spine) obtained by surgery from a number of AS patients 5,6. The presence of T cell and other MNC infiltrates was strongly dependent on the presence of cartilage on the surface of the femoral heads, suggesting that cartilage could be indeed the stimulus and target of a cellular immune response. Furthermore, T cell responses have been demonstrated against proteoglycan (an important cartilage protein) in human arthritides including ankylosing spondylitis . We could also recently demonstrate both a CD4+ and a CD8+ T cell response to proteoglycan (aggrecan) derived peptides in the peripheral blood and a CD8+ T cell response against a collagen VI derived peptide in the synovial fluid from AS patients. Thus, all these findings suggest that a chronic, probably T cell mediated, immune response against cartilage is relevant in the pathogenesis of AS.Further strong evidence for a crucial role of T cells in the pathogenesis of AS comes, in addition to the experimental data discussed above, from the association of AS with the MHC class I antigen HLA-B27. Because the natural function of HLA molecules is the presentation of peptides to T cells it has been postulated that the presentation of a yet unknown peptide to T cells might be the link to explain this HLA-B27 association , although direct evidence for this hypothesis is still missing. However, this hypothesis is backed by a lack of association with the HLA-B27 subtypes *B2706 and *B2709, which differ from the other susceptible subtypes by only 1 (or 2) amino acid substitution at the bottom of the peptide binding groove . Thus, these subtypes might not present an arthritogenic peptide. Based on the above described findings about the role of T-cells in ankylosing spondylitis we assume that Abatacept has the potential to be an effective drug for treating ankylosing spondylitis.The rheumatology group at the Charité, Campus Benjamin Franklin, has a large experience in the conduction of clinical trials, especially in ankylosing spondylitis, including treatment with biologicals . The infliximab trials finally led to the approval of infliximab for the indication ankylosing spondylitis. Most of these studies were conducted as investigators' initiated (sponsored) trials. From these trials we know that the placebo response rate is rather small in patients with active ankylosing spondylitis. The aim of the proposed trial is to evaluate the short-term efficacy and safety of treatment of active AS (BASDAI > 4 despite adequate therapy with NSAIDs) in a pilot open label trial with abatacept. If a clear response (see sample size justification). with an acceptable safety can be reached this study would be followed by a double blind placebo-controlled trial.We propose to treat in this open label pilot study two groups of patients: 1. TNFa-blocker failures (meaning patients who did not show an adequate response to TNFa-blocker treatment according to the international ASAS recommendations 7; not meaning patients who had to be discontinued because of side effects) and 2. TNFa-blocker naïve patients. We expect to gain important information about potential indications for treatment of AS with abatacept already by a relatively simple study design and a small number of patients (N= 30 in total).Research hypothesis The aim of the proposed trial is to evaluate the short-term efficacy and safety of treatment of active AS (BASDAI > 4 despite adequate therapy with NSAIDs) in a pilot open label trial with abatacept. If a clear response (see sample size justification) with an acceptable safety can be reached this study would be followed by a double blind placebo-controlled trial.

ELIGIBILITY:
Inclusion Criteria:

Patients 18 - 65 years of age who have moderate to severe ankylosing spondylitis.

1. Patients 18- 65 years of age who have moderate to severe ankylosing spondylitis.
2. Group

   1. TNFalpha inhibitor naïve patients: active AS patients with inadequate response to conventional therapy (e.g. NSAIDs, glucocorticosteroids or DMARDs) or with intolerance of conventional therapy Group
   2. TNFalpha inhibitor failures: active AS patients with inadaequate response to treatment with TNFalpha inhibitors (= patients with previous treatment with TNFalpha inhibitors who showed an inadaquate response according to the international ASAS recommendations; NOT AS patients who had to discontinue TNFalpha inhibitor treatment because of intolerance)
3. active disease is defined as a BASDAI score of>= 4, back pain score (BASDAI question 2) of >= 4 despite concurrent NSAID therapy, or intolerance to NSAIDs (first group) or prior treatment with TNFalpha inhibitors (second group)
4. if on NSAIDs, dosage must be stable 2 weeks prior to baseline. During the study dosage should be stable but is allowed to be reduced if documentated.
5. If on prednisone, <=10.0 mg per day, must be stable for 4 weeks prior to baseline and should be kept stable during the study
6. If on sulfasalazine or methotrexate, must be stable for 4 weeks prior to baseline
7. If on TNFalpha blocking agent (infliximab, etancercept, adalimumab), the TNFa therapy must have been terminated at least 4 weeks prior to baseline if etanercept was used and at least 8 weeks if infliximab or adalimumab were used.

Exclusion Criteria:

Main Inclusion/Exclusion Criteria

Exclusion criteria related to general health conditions

1. Current clinical or laboratory evidence of active or latent tuberculosis (TB) and subjects with a history of active TB treated within the last 3 years --> all potential subjects will have a screening chest x-ray at baseline (acceptable if present within the last 3 months); all potential subjects will have a Tuberculin skin test at screening
2. Patients with other chronic inflammatory articular disease or systemic autoimmune disease, e.g. Systemic lupus erythematosus, Sjögren's syndrome, active rheumatoid vasculitis, a history of systemic diseases associated with arthritis, chronic fatigue syndrome (other manifestations of spondyloarthritis such as psoriasis, inflammatory bowel disease, arthritis, uveitis are not regarded as exclusion criteria)
3. Any active infection, a history of recurrent clinically significant infection, a history of recurrent bacterial infections with encapsulated organisms
4. Hepatitis B or C or HIV
5. Primary or secondary immunodeficiency
6. History of cancer with curative treatment not longer than 5 years ago except basal-cell carcinoma of the skin that had been excised
7. A history of pulmonary or cardiac insufficiency, or serious and/or uncontrolled diseases that are likely to interfere with the evaluation of the patient's safety and of the study outcome
8. Evidence of significant uncontrolled concomitant diseases such as cardiovascular disease ( e.g. heart failure class III/IV NYHA, cardiac infarct within last 6 month), nervous system, pulmonary, renal, hepatic, endocrine or gastrointestinal disorders.
9. Neuropathy that can interfere with quality of life and/or pain assessment.
10. Patients with a history of a severe psychological illness or condition such as to interfere with the patient's ability to understand the requirements of the study.
11. History of current evidence of abuse of "hard" drugs (e.g. cocaine/ heroine) or alcoholism
12. Known hypersensitivity to any component of the study medication
13. Women lactating, pregnant, nursing or of childbearing potential with a positive pregnancy test (urine test)
14. Males or females of reproductive potential not willing to use effective contraception (e.g. contraceptive pill, IUD, physical barrier)
15. History of alcohol, drug or chemical abuse within 6 month prior to screening

Exclusion criteria related to medications

1. if previously on TNFalpha blocking agents, discontinuation of TNFalpha-blocking agents because of intolerance
2. If on leflunomide, leflunomide must have been terminated at least 8 weeks prior to the first abatacept administration (or ≥ 28 days after 11 days of standard cholestyramine or activated charcoal washout).
3. If on TNFalpha blocking agent (infliximab, etancercept, adalimumab), the TNFa therapy must have been terminated at least 4 weeks prior to the first abatacept adminstration if etanercept was used and at least 8 weeks if infliximab or adalimumab were used
4. Previous treatment with abatacept
5. If on sulfasalazine or methotrexate, must be stable for 4 weeks prior to baseline
6. Corticosteroids at doses exceeding 10 mg per day of prednisolone or the equivalent within the last 4 weeks prior to the first abatacept administration
7. Previous treatment with any investigational agent within 28 days ( or less than 5 terminal half-lives of elimination) of day 1 dose
8. Previous treatment with i.v. immunoglobulin
9. Receipt of a live vaccine within 4 weeks prior to treatment
10. Intra-articular or parenteral corticosteroids within 4 weeks prior to screening visit

Exclusion criteria related to lab findings

1. Haemoglobin < 8.5 g/dl
2. Neutrophil counts < 2.000 / µl
3. Platelet count < 125.000 / µl
4. Lower than 1 x 1000/µl lymphopenia for more than three months prior to inclusion.
5. Serum creatinine > 1.4 mg/dl for women or 1.6 mg/dl for men.
6. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2.5 times upper limit of normal
7. Positive HIV, hepatitis B or C serology
8. Any other laboratory test result that, in the opinion of the investigator, might place the subject at unacceptable risk for participation in this study.

Exclusion criteria related to formal aspects

1. Patients who participate currently in another clinical trial or patients who participated in another clinical trial during the last 30 days.
2. Patients who are underage or patients who are incapable to understand the aim, importance and consequences of the study and to give legal informed consent (according to § 40 Abs. 4 and § 41 Abs. 2 und Abs. 3 AMG).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-01; Primary Completion 2009-10; Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
ASAS40 response rate in TNF-blocker naïve and in TNF-blocker failure patients | at week 24

SECONDARY OUTCOMES:
Safety Evaluations: Adverse events, vital signs, physical examination results, and clinical laboratory values | until week 36
ASAS20 response | througout study
ASAS partial remission criteria | throughout study
BASDAI 20 response | throughout study
BASDAI 50 response | throughout study
BASFI | throughout study
BASMI | throughout study
C-reactive protein | throughout study
erythrocyte sedimentation rate | throughout study
Quality of Life: SF-36, AS-QoL, EQ-5D | Quality of Life: SF-36, AS-QoL, EQ-5D
Numeric Rating Scale (NRS) - physicians global, patients global, general pain, nocturnal pain | throughout the study
Enthesitis index (Maastricht scale) | throughout the study
swollen and tender joint count | swollen and tender joint count
Socio-economic questionnaire | throughout the study
course of change of active and chronic inflammatory lesions in MRI | throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Sieper, MD, Principal Investigator — Charité University Medicine Berlin, Campus Benjamin Franklin, Medical Department I, Rheumatology, Hindenburgdamm 30, 12200 Berlin, Germany
Locations (2):
- Germany (2):
  - Charité University Medicine Berlin, Campus Benjamin-Franklin, Berlin
  - Rheumazentrum Ruhrgebiet, Herne

REFERENCES:
- [Background] Zochling J, van der Heijde D, Burgos-Vargas R, Collantes E, Davis JC Jr, Dijkmans B, Dougados M, Geher P, Inman RD, Khan MA, Kvien TK, Leirisalo-Repo M, Olivieri I, Pavelka K, Sieper J, Stucki G, Sturrock RD, van der Linden S, Wendling D, Bohm H, van Royen BJ, Braun J; 'ASsessment in AS' international working group; European League Against Rheumatism. ASAS/EULAR recommendations for the management of ankylosing spondylitis. Ann Rheum Dis. 2006 Apr;65(4):442-52. doi: 10.1136/ard.2005.041137. Epub 2005 Aug 26. PMID 16126791
- [Background] Appel H, Kuhne M, Spiekermann S, Ebhardt H, Grozdanovic Z, Kohler D, Dreimann M, Hempfing A, Rudwaleit M, Stein H, Metz-Stavenhagen P, Sieper J, Loddenkemper C. Immunohistologic analysis of zygapophyseal joints in patients with ankylosing spondylitis. Arthritis Rheum. 2006 Sep;54(9):2845-51. doi: 10.1002/art.22060. PMID 16947385
- [Background] Appel H, Loddenkemper C, Grozdanovic Z, Ebhardt H, Dreimann M, Hempfing A, Stein H, Metz-Stavenhagen P, Rudwaleit M, Sieper J. Correlation of histopathological findings and magnetic resonance imaging in the spine of patients with ankylosing spondylitis. Arthritis Res Ther. 2006;8(5):R143. doi: 10.1186/ar2035. PMID 16925803
- [Background] Appel H, Kuhne M, Spiekermann S, Kohler D, Zacher J, Stein H, Sieper J, Loddenkemper C. Immunohistochemical analysis of hip arthritis in ankylosing spondylitis: evaluation of the bone-cartilage interface and subchondral bone marrow. Arthritis Rheum. 2006 Jun;54(6):1805-13. doi: 10.1002/art.21907. PMID 16736521
- [Background] Sieper J, Braun J. Pathogenesis of spondylarthropathies. Persistent bacterial antigen, autoimmunity, or both? Arthritis Rheum. 1995 Nov;38(11):1547-54. doi: 10.1002/art.1780381105. PMID 7488274
- [Background] Maksymowych WP. Ankylosing spondylitis--at the interface of bone and cartilage. J Rheumatol. 2000 Oct;27(10):2295-301. No abstract available. PMID 11036819
- [Background] Weinblatt M, Combe B, Covucci A, Aranda R, Becker JC, Keystone E. Safety of the selective costimulation modulator abatacept in rheumatoid arthritis patients receiving background biologic and nonbiologic disease-modifying antirheumatic drugs: A one-year randomized, placebo-controlled study. Arthritis Rheum. 2006 Sep;54(9):2807-16. doi: 10.1002/art.22070. PMID 16947384
- [Background] Kremer JM, Genant HK, Moreland LW, Russell AS, Emery P, Abud-Mendoza C, Szechinski J, Li T, Ge Z, Becker JC, Westhovens R. Effects of abatacept in patients with methotrexate-resistant active rheumatoid arthritis: a randomized trial. Ann Intern Med. 2006 Jun 20;144(12):865-76. doi: 10.7326/0003-4819-144-12-200606200-00003. PMID 16785475